CLINICAL TRIAL: NCT00223652
Title: Tele-Mental Health Intervention to Improve Depression Outcomes in Community Based Outpatient Clinics (CBOCs)
Brief Title: Telephone Administered Psychotherapy for the Treatment of Depression for Veterans in Rural Areas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 03-069
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-08

CONDITIONS: Depressive Disorder; Depression
Keywords: Cognitive-Behavioral Therapy; Telephone psychotherapy; Clinical Trial; Primary Care Clinic; Treatment for Depression
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 - Telephone CBT (Experimental): Telephone cognitive behavioral therapy
  Interventions: Behavioral: Telephone cognitive behavioral therapy
- Arm 2 - Treatment as Usual (No Intervention): Treatment as usual control.

INTERVENTIONS:
Behavioral: Telephone cognitive behavioral therapy — An initial treatment phase consisting of 12 weekly sessions aimed at reducing symptoms of depression, and a booster phase in which 4 sessions are provided at increasingly greater intervals to target maintenance of treatment gains.
  Arms: Arm 1 - Telephone CBT

SUMMARY:
The purpose of this study is to examine the efficacy of telephone-administered cognitive-behavioral therapy (T-CBT) in treating major depression among veterans served by community-based outpatient clinics (CBOCs) in the Veteran's Integrated Service Network (VISN) 21, which serves rural areas in Northern California and (VISN) 12, which serves rural areas surrounding the Hines, IL VA Hospital.

DETAILED DESCRIPTION:
More than 20% of patients in primary care have depressive disorders. While primary care is the principal venue for treatment for depression, fewer than 25% of depressed patients receive adequate treatment for their depression. These outcomes can be worse when there are barriers to treatment such as living in a rural area. Several studies have found that given a choice, about two-thirds of depressed primary care patients prefer psychotherapy or counseling over antidepressant medication.

This is a controlled, randomized trial in which subjects meeting criteria for major depressive disorder (MDD) from primary care settings in VISN 21 including CBOCs will be randomly assigned to one of two conditions: 1) a 16-session manualized telephone administered cognitive behavioral therapy (T-CBT) delivered over 20 weeks or 2) a treatment-as-usual (TAU) condition. Telephone-administered cognitive behavioral therapy (T-CBT) is an intervention aimed at improving coping skills and social functioning. It is divided into two phases: 1) an initial treatment phase consisting of 12 weekly sessions aimed at reducing symptoms of depression, and 2) a booster phase in which 4 sessions are provided at increasingly greater intervals to target maintenance of treatment gains. T-CBT, administered by doctoral level psychologists, will be compared to a treatment-as-usual (TAU) condition that controls for the natural course of depression during the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has a DSM-IV diagnosis of Major Depressive Disorder as assessed using the MINI
* Has a telephone
* Able to speak and read English
* At least 18 years of age
* Able to give informed consent
* Must be registered at a VA community-based, outpatient clinic (CBOC) at VA Eureka or VA Ukiah or VA Santa Rosa, or VA Manteno, or VA Elgin, or VA La Salle

Exclusion Criteria:

* Has a hearing, voice or visual impairment that would prevent participation in T-CBT
* Meets criteria for dementia
* Is diagnosed with Psychotic Disorder, Bipolar Disorder, substance abuse with clinical consensus, or current severe PTSD.
* Is currently receiving psychotherapy or planning to receive psychotherapy during the 20-week treatment phase of the study
* Has a history of suicide attempts or is at high risk for suicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2006-03; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C. Mohr, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois

REFERENCES:
- [Result] Mohr DC, Vella L, Hart S, Heckman T, Simon G. The Effect of Telephone-Administered Psychotherapy on Symptoms of Depression and Attrition: A Meta-Analysis. Clin Psychol (New York). 2008;15(3):243-253. doi: 10.1111/j.1468-2850.2008.00134.x. PMID 21369344
- [Result] Mohr DC, Carmody T, Erickson L, Jin L, Leader J. Telephone-administered cognitive behavioral therapy for veterans served by community-based outpatient clinics. J Consult Clin Psychol. 2011 Apr;79(2):261-5. doi: 10.1037/a0022395. PMID 21299274

RESULTS

PARTICIPANT FLOW:
Groups:
- Telephone-administered Cognitive-Behavioral Therapy: Telephone cognitive behavioral therapy
  Telephone-administered Cognitive-Behavioral Therapy (T-CBT): An initial treatment phase consisting of 12 weekly sessions aimed at reducing symptoms of depression, and a booster phase in which 4 sessions are provided at increasingly greater intervals to target maintenance of treatment gains.
- Treatment as Usual: Treatment as usual control.
Period: T-CBT 12 Weeks, TAU 20 Weeks
Arm/Group | Telephone-administered Cognitive-Behavioral Therapy | Treatment as Usual
Started | 41 | 44
Completed | 40 | 41
Not Completed | 1 | 3
Period: T-CBT 20 Weeks, TAU 20 Weeks
Arm/Group | Telephone-administered Cognitive-Behavioral Therapy | Treatment as Usual
Started | 40 | 41
Completed | 40 | 41
Not Completed | 0 | 0
Period: T-CBT and TAU 6 Month Follow-up
Arm/Group | Telephone-administered Cognitive-Behavioral Therapy | Treatment as Usual
Started | 40 | 41
Completed | 39 | 37
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone-administered Cognitive-Behavioral Therapy | Treatment as Usual | Total
Number analyzed (Participants) | 41 | 44 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.83 (10.81) | 54.98 (10.42) | 55.9 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 38 | 39 | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 33 | 34 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 41 | 44 | 85

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Depression Using Hamilton Depression Rating Scale
Description: Evaluators administered the Hamilton Depression Rating Scale(Ham-D).
  Veterans were assessed at baseline,12 weeks, 20 weeks(posttreatment), and 6-month follow-up using the Ham-D. Self-reported depression was measured using the Hamilton Depression Rating Scale(Ham-D).
  Data across the three time points (baseline, Week 12, Week 20) were analyzed using a mixed-effects repeated measures model with random subject-specific intercepts for continuous outcome Ham-D.
  Ham-D ranges from 0-52, higher values indicate more severe depression. A score of 0-7 is considered to be normal. Scores of 20 or higher indicate moderate, severe, or very severe depression.
Time Frame: Baseline, 12 weeks, 20 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone-administered Cognitive-Behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 41 | 44
units on a scale
  Baseline, n = 41, n = 44, respectively | 20.83 (3.96) | 19.23 (3.72)
  Week 12, n = 40, n = 41 respectively | 16.71 (6.42) | 17.27 (5.29)
  Week 20, n = 40, n =41, respectively | 15.43 (5.51) | 17.00 (5.68)
Statistical Analysis 1: Comparison: Telephone-administered Cognitive-Behavioral Therapy vs Treatment as Usual; Test type: Superiority or Other; p = .001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Telephone-administered Cognitive-Behavioral Therapy vs Treatment as Usual; Test type: Superiority or Other; p = 0.07, Mixed Models Analysis
Statistical Analysis 3: Comparison: Telephone-administered Cognitive-Behavioral Therapy vs Treatment as Usual; Test type: Superiority or Other; p = 0.95, Mixed Models Analysis

2. Secondary Outcome: Maintenance of Treatment Effect
Description: Evaluators administered the Hamilton Depression Rating Scale(Ham-D). Veterans were assessed at baseline,12 weeks, 20 weeks(post treatment), and 6-month follow-up using the Ham-D.Data was analyzed using a mixed-effects repeated measures model with random subject-specific intercepts for continuous outcome Ham-D.
  Ham-D ranges from 0-52, higher values indicate more severe depression. A score of 0-7 is considered to be normal. Scores of 20 or higher indicate moderate, severe, or very severe depression.
Time Frame: 6 month follow-up (week 44)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone-administered Cognitive-Behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 39 | 37
units on a scale | 13.62 (6.36) | 14.81 (5.01)
Statistical Analysis 1: Comparison: Telephone-administered Cognitive-Behavioral Therapy vs Treatment as Usual; Test type: Superiority or Other; p > 0.37, Mixed Models Analysis

3. Primary Outcome: Change in Severity of Depression Using the Patient Health Questionnaire-9
Description: Self-reported depression was measured using the Patient Health Questionnaire-9 (PHQ-9).
  Data across the three time points (baseline, Week 12, Week 20) were analyzed using a mixed-effects repeated measures model with random subject-specific intercepts for continuous outcome PHQ-9. PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe and severe depression, respectively.
  PHQ-9 score ranges from 0-27, higher values indicate more severe depression.
Time Frame: Baseline, Week 12, Week 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Telephone-administered Cognitive-Behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 41 | 44
units on a scale
  Baseline, n = 41, n = 44, respectively | 17.12 (5.10) | 17.39 (4.79)
  Week 12, n = 40, n = 41, respectively | 12.19 (5.96) | 14.35 (6.05)
  Week 20, n = 40, n = 41, respectively | 11.15 (6.46) | 12.90 (5.28)
Statistical Analysis 1: Comparison: Telephone-administered Cognitive-Behavioral Therapy vs Treatment as Usual; Test type: Superiority or Other; p < .0001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Telephone-administered Cognitive-Behavioral Therapy vs Treatment as Usual; Test type: Superiority or Other; p = 0.61, Mixed Models Analysis
Statistical Analysis 3: Comparison: Telephone-administered Cognitive-Behavioral Therapy vs Treatment as Usual; Test type: Superiority or Other; p = 0.20, Mixed Models Analysis

4. Primary Outcome: Number of Participants Meeting Criteria for Major Depressive Disorder
Description: Veterans meeting criteria for major depressive disorder were randomized to receive 16 session of T-CBT over 20 weeks or treatment as usual through the CBOC. Generalized estimating equations models with exchangeable working correlation structure was used for the binary outcome (MDE). A veteran was required to meet diagnostic criteria for severe psychiatric disorder(e.g., psychotic, bipolar, or dementia disorder; post-traumatic stress disorder [PTSD] patients were not excluded). DSM-IV diagnosis was assessed using the full Mini International Neuropsychiatric Interview at baseline, whereas the major depressive episode(MDE) module was administered at follow-up.
Time Frame: Baseline to week 12, and week 20
Measure: Number; unit: participants
Arm/Group | Telephone-administered Cognitive-Behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 41 | 44
participants
  number of particpants with MDE at Baseline | 41 | 44
  number of particpants with MDE Week 12 | 20 | 29
  number of particpants with MDE Week 20 | 19 | 23
Statistical Analysis 1: Comparison: Telephone-administered Cognitive-Behavioral Therapy vs Treatment as Usual; Test type: Superiority or Other; p < 0.0001, Generalized estimating equations models
Statistical Analysis 2: Comparison: Telephone-administered Cognitive-Behavioral Therapy vs Treatment as Usual; Test type: Superiority or Other; p = 0.12, Generalized estimating equations models
Statistical Analysis 3: Comparison: Telephone-administered Cognitive-Behavioral Therapy vs Treatment as Usual; Test type: Superiority or Other; p = 0.86, Generalized estimating equations models

5. Secondary Outcome: Maintenance of Treatment Effect
Description: 6-month post treatment follow-up on outcome measure of the Patient Health Questionnaire-9 (PHQ-9).
  Data was analyzed using a mixed-effects repeated measures model with random subject-specific intercepts for continuous outcome PHQ-9.
  PHQ-9 score ranges from 0-27, higher values indicate more severe depression. PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe and severe depression, respectively.
Time Frame: 6-month post treatment follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Telephone Cognitive Behavioral Therapy: Telephone cognitive behavioral therapy
  Telephone-administered Cognitive-Behavioral Therapy (T-CBT): An initial treatment phase consisting of 12 weekly sessions aimed at reducing symptoms of depression, and a booster phase in which 4 sessions are provided at increasingly greater intervals to target maintenance of treatment gains.
Arm/Group | Telephone Cognitive Behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 39 | 37
units on a scale | 11.25 (6.67) | 12.26 (5.63)
Statistical Analysis 1: Comparison: Telephone Cognitive Behavioral Therapy vs Treatment as Usual; Test type: Superiority or Other; p > 0.37, Mixed Models Analysis

6. Secondary Outcome: Number of Participants Meeting Criteria for Major Depression Disorder at 6 Month Follow-up
Description: as for outcome 4
Time Frame: 6-month follow up at week 44 post treatment
Measure: Number; unit: participants
Arm/Group | Telephone Cognitive Behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 39 | 37
participants | 16 | 18
Statistical Analysis 1: Comparison: Telephone Cognitive Behavioral Therapy vs Treatment as Usual; Test type: Superiority or Other; p > 0.37, Generalized estimating equations models

ADVERSE EVENTS:
Arm/Group | Telephone-administered Cognitive-Behavioral Therapy | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/44
Other Adverse Events (participants affected / at risk) | 0/41 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No